CLINICAL TRIAL: NCT02523222
Title: Prophylactic Dextrose Gel Does Not Prevent Neonatal Hypoglycemia: a Quasi-experimental Pilot Study
Brief Title: Dextrose Gel Does Not Prevent Neonatal Hypoglycemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohan Pammi, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-36132
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Hypoglycemia; Infant, Small for Gestational Age; Premature Birth of Newborn; Fetal Macrosomia; Intrauterine Growth Restriction; Complication of Prematurity; Neonatal Hypoglycemia
Keywords: dextrose gel; newborn hypoglycemia; late preterm infant; large for gestational age; small for gestational age; prophylactic; neonatal hypoglycemia
MeSH Terms: conditions — Hypoglycemia; Premature Birth; Fetal Macrosomia; Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL (No Intervention): Infants at risk for transient neonatal hypoglycemia following standard-of-care.
- Dextrose Gel (Active Comparator): Infants given 40% Dextrose gel (0.5ml/kg) in the buccal mucosa after their first feed, within the first hour of life.
  Interventions: Dietary Supplement: 40% Dextrose gel

INTERVENTIONS:
Dietary Supplement: 40% Dextrose gel — 40% dextrose gel will be rubbed into the hypoglycemic infant's buccal mucosa at a dose of 0.5ml/kg.
  Arms: Dextrose Gel

SUMMARY:
This was a quasi-experimental pilot study comparing blood glucose values 30 minutes after feeding alone or feeding + dextrose gel in newborns at risk for transient neonatal hypoglycemia.

DETAILED DESCRIPTION:
OBJECTIVE: To test the hypothesis that prophylactic dextrose gel administered to newborns at risk for hypoglycemia will increase the initial blood glucose (BG) concentration after the first feeding and subsequently decrease NICU admissions for treatment of asymptomatic transient neonatal hypoglycemia (TNH) vs those given feedings alone.

STUDY DESIGN: This quasi-experimental pilot study allocated asymptomatic at-risk newborns (late preterm, birth weight <2500 or >4000 g, and infants of diabetic mothers) to receive prophylactic dextrose gel (Insta-Glucose®); other at-risk newborns served as controls. After the initial feeding, the prophylactic group received dextrose gel (0.5 ml/kg) rubbed into the buccal mucosa, and BG was checked 30 min later. Initial BG concentrations and rate of NICU admissions (for treatment of hypoglycemia) were compared between the prophylactic group and controls using the Wilcoxon rank-sum test and Fisher's exact test, where appropriate. A multivariable linear regression compared first BG between groups after adjusting for at-risk categories and age at first BG concentration.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age above 35 weeks
* Infants less than 1 hour of age
* Infants with informed parental consent
* Infants who are born at the Harris Health Ben Taub Hospital in Houston, TX

Exclusion Criteria:

* Infants with known metabolic, genetic, or congenital anomalies
* Infants not expected to survive the neonatal period
* Infants determined later to have a metabolic, genetic, or congenital anomaly that was not immediately obvious in the newborn period
* Hypoglycemic infants with symptoms
* Infants transferred to the Level 3 NICU for other reasons

Ages: 0 Hours to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Prophylactic administration of dextrose gel | 2 hours
  Give infants who meet criteria for high-risk and whose parents have consented one dose of prophylactic 40% dextrose gel (0.5ml/kg) after first feed. Assess glucose level after 1 feed and 1 application of dextrose gel, and admission to the NICU, compared to controls with similar risk factors who are not treated prophylactically.
Treatment failure of at-risk infants | 4 days
  Infants at-risk (IDM, late preterm, SGA, LGA, estimated fetal weight below 2.5kg or above 4kg, IUGR, or poor feeding) will be followed until hospital discharge to measure NICU admission data and glucose values during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Kaiser, MD, MA, FAAP, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Ben Taub Harris Health Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coors SM, Cousin JJ, Hagan JL, Kaiser JR. Prophylactic Dextrose Gel Does Not Prevent Neonatal Hypoglycemia: A Quasi-Experimental Pilot Study. J Pediatr. 2018 Jul;198:156-161. doi: 10.1016/j.jpeds.2018.02.025. Epub 2018 Mar 28. PMID 29605395